CLINICAL TRIAL: NCT01249092
Title: A Pilot Study of Pentoxifylline for the Treatment of Primary Biliary Cirrhosis
Brief Title: Pentoxifylline for Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Claudia Zein, MD, Staff Physician, Digestive Disease Institute, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-1003
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-10

CONDITIONS: Primary Biliary Cirrhosis
Keywords: biliary cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pentoxifylline 400 mg TID (Experimental): This study is an open label pilot with only one arm.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Patients will take 400mg of pentoxifylline three times daily for a total duration of 6 months.

SUMMARY:
Primary biliary cirrhosis (PBC) is cholestatic liver disease characterized by progressive destruction of small bile ducts within the liver that can lead to end stage liver disease and all its complications.

Although ursodeoxycholic acid (UDCA) is associated with increased survival in many patients with PBC, there is absence of an adequate response to UDCA in a significant proportion of PBC patients.

Tumor necrosis factor alpha (TNF-alpha) is a cytokine that plays an important role in the pathogenesis of PBC. Other fibrosis biomarkers such as tissue metallo proteinase 1 (TIMP-1) are associated with progression of liver fibrosis in PBC. Pentoxifylline (PTX) is a methylxanthine derivative that inhibits pro-inflammatory cytokines and also has shown anti-fibrotic effects in serum of patients with PBC. Furthermore, PTX has well known clinical and safety profiles. The main hypothesis of this study is that therapy with pentoxifylline (PTX) will result in improvement of liver disease in PBC patients who are incomplete responders to UDCA.

The focus of this proposal is on the effectiveness of PTX in improving laboratory parameters of liver disease and levels of cytokines involved in the pathogenesis of the disease in patients with PBC.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18 to 76 years.
* Established diagnosis of PBC based on at least three of the following criteria:

  * Detectable anti-mitochondrial antibodies (AMA)
  * Cholestatic biochemical pattern
  * Liver biopsy compatible with PBC
  * Appropriate exclusion of other liver diseases.
* Therapy with UDCA at adequate dose (13-15mg/kg/d) for at least six months and evidence of suboptimal response defined by alkaline phosphatase levels that did not normalize and remain elevated by at least 1.5 times the upper limit of normal.
* No history or present hepatic decompensation (e.g. variceal hemorrhage, encephalopathy, or poorly controlled ascites).

Exclusion Criteria:

* Findings highly suggestive of liver disease of other etiology.
* A score >=10 points on the Revised Scoring System for autoimmune hepatitis (AIH), supporting a diagnosis of PBC/AIH overlap.
* Patients on steroids (systemic), immunosuppressants, or immunomodulatory agents within the previous 6 months.
* Patients with clinical or laboratory evidence suggestive of decompensated cirrhosis.
* Hypersensitivity to PTX or the methylxanthines (caffeine, theophylline, theobromine).
* History of cerebral or retinal hemorrhage.
* Other medical comorbidities (such as cardiac, renal, cancer) that would interfere with completion of the study.
* Patients taking Theophylline or Coumadin because of potential drug-drug interactions with PTX. In addition, patients taking low molecular weight heparin preparations.
* Pregnant or nursing women.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia O. Zein, MD, MSc, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment was initiated in December 2010 and a total of 20 patients were enrolled. The last patient to complete the pilot study completed participation in June 2012.
Pre-assignment Details: This was a single arm open label pilot study where all subjects received the same intervention throughout the study duration. There were no different study groups and no randomization was involved.
Groups:
- Pentoxifylline 400 mg/d: All patients received same intervention.
Period: Overall Study
Arm/Group | Pentoxifylline 400 mg/d
Started | 20
Completed | 18
Not Completed | 2
Not completed — Expected side effect of nausea/dyspepsia | 1
Not completed — Unable to tolerate expected SE -nausea | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pentoxifylline 400 mg/d
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 57.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Alkaline Phosphatase Levels.
Description: Serum alkaline phosphatase levels at entry and at 6 months of therapy with PTX will be measured and compared.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Change in Alkaline Phosphatase After Pentoxifylline Therapy
Number analyzed (Participants) | 18
U/L | -57.3 (62.1)
Statistical Analysis 1: Comparison: Change in Alkaline Phosphatase After Pentoxifylline Therapy; A p-value < 0.05 was considered statistically significant and all analyses were carried out using SAS version 9.2 (The SAS Institute, Cary, NC). Matched pairs t-test was used to compare the change in alkaline phosphatase from baseline. The efficacy of therapy was measured based on improvement in AP levels after therapy with PTX. AP levels at end of the study were compared with values at baseline by matched pairs t-test; Test type: Superiority or Other; p = 0.001, Paired t-test — This study tested the hypothesis that treatment with pentoxifylline would result in a statistically significant change from baseline in the level of alkaline phosphatase; Mean Difference (Final Values) = -57.3, 95% CI 2-sided [-88.2 to -26.4], Standard Deviation 62.1

2. Secondary Outcome: Change in Serum Concentration of Tissue Inhibitor Metalloproteinase 1 (TIMP-1) After PTX Therapy.
Description: Serum concentration of tissue inhibitor metalloproteinase 1 (TIMP-1), a fibrosis biomarker of interest, will be measured and the change in serum levels between entry and end of study will be calculated.
Time Frame: 6 months
Population: Serum samples from both timepoints (entry and end of study) were available in only 16 of the 18 subjects who completed the study.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Change in Serum TIMP-1 (Tissue Inhibitor metalloproteinase1)
Number analyzed (Participants) | 16
ng/mL | -5.69 (8.66)
Statistical Analysis 1: Comparison: Change in Serum TIMP-1 (Tissue Inhibitor metalloproteinase1); Change from baseline in TIMP-1 levels was assessed by paired-t test. Distribution the variable values was assessed using normal probability plots. Matched pairs t-test was used to compare the change from baseline; Test type: Superiority or Other; p = 0.5, Paired t-test. — Hypothesis tested if TIMP-1 levels after therapy with pentoxifylline changed significantly from baseline from baseline; Mean Difference (Net) = -5.69, 95% CI 2-sided [-24.14 to 8.68], Standard Error of Mean 8.66

3. Secondary Outcome: Safety of Therapy in the Pilot Study of PTX Therapy in Patients With PBC Will be Assessed
Description: The number of participants that experienced any severe adverse events will be monitored and recorded.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Pentoxifylline 400 mg/d: Descriptive information only of small open label pilot. Small patient number not amenable for any valid statistical comparisons regarding side effects. All patients received same intervention. No SAEs occurred.
Arm/Group | Pentoxifylline 400 mg/d
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: 2 years and 6 months
Description: Patients were followed for adverse events and side effect through the duration of the study and on subsequent follow up. Patients were contacted directly by PI and questionnaire about adverse effects was completed at weeks 4, 8, 12, 16, 20, and 24 during the study and then subsequently on follow up.
Arm/Group | Pentoxifylline 400 mg/d
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline 400 mg/d (N=20)
Nausea (Gastrointestinal disorders) | 7 (7) — Nausea rated more than mild temporary nausea (mild temporary nausea commonly occurs for a few days when initiating pentoxifylline)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Our study was a small open label pilot completed with no technical problems. The information generated will be useful in designing future larger studies. The main limitation is that PBC is a rare disease which resulted in prolonged enrollment phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No